CLINICAL TRIAL: NCT03284307
Title: UNderstanding CONSciousness Connectedness and Intraoperative Unresponsiveness Study
Acronym: UN-CONSCIOUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-1399; A530900 (Other: UW Madison); SMPH\ANESTHESIOLOGY\ANESTHESIO (Other: UW Madison); Protocol Version 10/18/2019 (Other: UW Madison)
Record Dates: First submitted 2017-08-22; First posted 2017-09-15 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Unconsciousness; Consciousness
Keywords: Sedation; Propofol; Dexmedetomidine; Ketamine; Sevoflurane; Electroencephalogram
MeSH Terms: conditions — Unconsciousness | interventions — Dexmedetomidine; Ketamine; Propofol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Drug Administrated (Experimental): Sedatives will be administered to participants while their brain activity is measured.
  Interventions: Drug: Dexmedetomidine; Drug: Ketamine; Drug: Propofol; Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — 20 participants will be administered Dexmedetomidine.
Drug: Ketamine — 20 participants will be administered Ketamine.
Drug: Propofol — 20 participants will be administered Propofol.
Drug: Midazolam — 20 participants will be administered Midazolam.

SUMMARY:
This study will be a single-site, controlled, unblinded study at the University of Wisconsin to examine changes in the electroencephalogram during anesthesia and waking.

DETAILED DESCRIPTION:
* 20 subjects will be recruited per drug, and subjects can be recruited to undergo multiple sedation protocols.

Screening:

Subjects will respond to the volunteer posts for the study by calling into a study specific phone number. They will complete a phone screening to determine basic eligibility for the study. At the beginning of the sedation session, participants will affirm that in the interval since their baseline visit, they have not acquired any of the cited exclusion criteria that would preclude participation. A review of these exclusion criteria will be completed by the Anesthesiologist. A standard pre-anesthetic assessment will be performed, including confirmation of NPO status, and documented using the standard Department of Anesthesiology pre-operative evaluation form.

The first sedative will be dexmedetomidine followed by ketamine, propofol and then midazolam (dependent on the availability of the drugs). Total enrollment in the study will be up to 80 subjects. Each sedation experiment will occur on separate days at least 28 days apart, if the subject chooses to participate in more than one session.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* In good health, determined by the PI on the basis of medical history and a standard assessment for anesthesia to be documented as part of the study record
* Right handed, to standardize for asymmetry in brain functions

Exclusion Criteria:

* Adults <18 years old or >40 years old
* Pregnancy confirmed on pregnancy test on day of sedation
* Contraindication to anesthesia or allergy to study drug
* Difficult anesthesia: American Society of Anesthesiologists Physical Status greater than 1, per the discretion of the PI. Examples of ASA status include, but are not limited to:

  * Any systemic disease present, such as diabetes, cardiac, pulmonary, or other acute or chronic disorder, or history of smoking
  * Narrow angle glaucoma
  * Abnormal airway examination
  * Any abnormality on medical history and physical examination
  * Snoring or sleep disorders including apnea
  * Antecedent pulmonary aspiration risk (e.g., history GI reflux, heartburn, hiatal hernia)
  * Adverse reaction or allergy with anesthesia or other sedatives
  * Chronic medication use
  * History of difficult anesthesia, laryngoscopy or intubation
  * Family history of difficulty with anesthesia or sedation
  * History of vertigo, nausea or vomiting after anesthesia
* BMI > 35
* Contraindication to HD-EEG, TMS or MRI for relative parts of the procedures. MRI exclusion criteria: presence of metallic or electronic implants; history of claustrophobia. TMS exclusion criteria: Presence or history of medical conditions that could increase the chance of seizures (e.g. - stroke, aneurysm, brain surgery, structural brain lesion) cranial metal implants; structural brain lesion; devices that may be affected by TMS (pacemaker, medication pump, cochlear implant, implanted brain stimulator); history of head trauma with loss of consciousness for greater than 5 minutes; family history of seizures; history of antecedent mood disorder.
* Exclusion from Dexmedetomidine:

  o Resting heart Rate<60 bpm
* Exclusion from Propofol:

  o Reported egg allergy
* Exclusion from Ketamine:

  * History of post-operative nausea and vomiting
  * History of motion sickness

Additional exclusion criteria on the day of sedation:

* Anything to eat or drink for the preceding 8 hours
* Any use of over-the-counter or recreational drugs (including alcohol or tobacco) within the preceding 24 hours
* Any use of sedative or sleep agents within the preceding 24 hours
* Recent change in health, including cough, cold, or fever
* Exposure to anesthesia or sedation in the last 6 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Pearce, MD, PhD, Principal Investigator — Professor and chair of Anesthesiology at UW- Madison
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Wehrman JJ, Casey C, Redinbaugh MJ, Muller E, Munn B, Payne T, Tanabe S, Mohanta S, Filbey W, Raz A, Banks MI, Pearce RA, Shine JM, Saalmann YB, Sanders RD. Thalamic contributions to predictive coding and disconnected consciousness in human volunteers. Br J Anaesth. 2025 Nov 27:S0007-0912(25)00776-7. doi: 10.1016/j.bja.2025.10.038. Online ahead of print. PMID 41314941
- [Derived] Casey CP, Tanabe S, Farahbakhsh ZZ, Parker M, Bo A, White M, Ballweg T, Mcintosh A, Filbey W, Banks MI, Saalmann YB, Pearce RA, Sanders RD. Evaluation of putative signatures of consciousness using specific definitions of responsiveness, connectedness, and consciousness. Br J Anaesth. 2024 Feb;132(2):300-311. doi: 10.1016/j.bja.2023.09.031. Epub 2023 Oct 31. PMID 37914581
- [Derived] Wehrman JJ, Casey C, Tanabe S, Mohanta S, Filbey W, Weber L, Banks MI, Pearce RA, Saalmann Y, Sanders RD. Subanaesthetic doses of ketamine reduce but do not eliminate predictive coding responses: implications for mechanisms of sensory disconnection. Br J Anaesth. 2023 Oct;131(4):705-714. doi: 10.1016/j.bja.2023.06.044. Epub 2023 Aug 3. PMID 37541951
- [Derived] Casey CP, Tanabe S, Farahbakhsh Z, Parker M, Bo A, White M, Ballweg T, Mcintosh A, Filbey W, Saalmann Y, Pearce RA, Sanders RD. Distinct EEG signatures differentiate unconsciousness and disconnection during anaesthesia and sleep. Br J Anaesth. 2022 Jun;128(6):1006-1018. doi: 10.1016/j.bja.2022.01.010. Epub 2022 Feb 9. PMID 35148892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via an email that was sent to UW-Madison students and staff from August 2017 through March 2020. Interested participants would discuss study commitment and preliminary screening criteria with the study team over the phone. Eligible participants would meet with a faculty anesthesiologist at a screening visit to complete informed consent and for a history and physical examination and basic neuropsychological assessment to determine subsequent study visit eligibility.
Pre-assignment Details: Participants were assigned to a drug if they were both eligible and reconsented the morning of the visit. Drug visits occurred in a sequence: Dexmedetomidine, Ketamine, Propofol, and then Midazolam. The same participant could participate in all drug visits if they were eligible, and a minimum of 28 days had past since their previous drug visit. All participants interested in a drug visit were asked to also complete a sleep visit which occurred before the first drug visit if possible.
Groups:
- All Study Participants: Participants completed sedation visits in the order of dexmedetomidine, ketamine, propofol, and midazolam. There was a washout period of at least 28 days between sedation visits. Subjects were also asked to complete a separate overnight sleep visit with an EEG. Participants reconsented at each sleep and sedation visit. If a patient was inappropriate for one sedative, due to a specific contraindication to that drug (and not the study in general) but were eligible for another drug, then they progressed through the order of sedatives while skipping that inappropriate drug.
  At each drug visit, participants were fitted with a saline gel EEG cap and a pre-sedation recording was collected. Participants' brain waves were recorded during rest, while responding to a standardized wake report form, and while performing a predictive coding cognitive task on a computer. Once the pre-sedation recording was collected, the faculty anesthesiologist began administering the study drug. A new EEG recording was started to monitor brain waves while all of the pre-sedation activities were repeated after the administration of the study drug.
Period: Overall Study
Arm/Group | All Study Participants
Started | 35
Completed Sedation and/or Sleep Visit | 27
Completed Sedation Visit | 21
Sleep (Participants were fitted with a saline gel EEG cap and a pre-sleep recording was collected. After the pre-sleep recording, participants laid down within 30 minutes of their usual bedtime and were left to sleep for 2-3 hours. Then, the participant was woken up every 15-30 minutes to answer standardized wake report form questions. After awaking a final time, the participant repeated 10 minutes of awake eyes open and eyes closed recordings and a predictive coding cognitive task on a computer.) | 15
Dexmedetomidine (Rapid infusion of 3.0 mg kg-1 h-1 was administered over a 10 min period followed by a 0.5 mg kg-1 h-1 maintenance infusion to achieve the first drug step. The second drug step was similarly achieved by a 10 min infusion of 3.0 mg kg-1 h-1 followed by a 1.5 mg kg-1 h-1 maintenance infusion. Duration of drug exposure was limited to 4 hours.) | 20
Ketamine (Ketamine was titrated using up to a 4.5mg/kg bolus over 10 minutes followed by 0.1-0.5mg/min intravenous infusion with 5 minutes between increments and titrated to desired observed alertness/sedation level. Short-lived emergence delirium (confusion on awakening) may occur on emergence from ketamine anesthesia and this will be managed through standard clinical practice including administration of midazolam (up to 4mg IV) if required. Duration of drug exposure was limited to 4 hours.) | 15
Propofol (A target-controlled infusion model used to predict plasma concentrations of propofol at 0.5 mcg/mL increments allowing 5-minutes to equilibrate between any step change. Dosing will be confined to FDA approved limits with up to a 2.5mg/kg bolus over 1 to 3 minute followed by an infusion of 50-200mcg/kg/min titrated to the desired observed alertness/sedation levels. Drug exposure was limited to 4 hours.) | 6
Midazolam (Initial boluses of up to 0.35mg/kg followed by doses up to 0.1mg/kg/h as a maintenance infusion. Duration of drug exposure was limited to 4 hours.) | 0 (No midazolam visit was ever conducted because no interested participants had reached that step of the drug sequence after it was added to the protocol in November of 2019.This was in large part due to the shutdown of in-person research activities in March of 2020 from the COVID-19 pandemic.)
Completed | 27
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: All participants who completed a sleep and/or sedation visit.
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed for each row is the number of participants who completed that visit.
  years
    Total | 23.44 (4.60)
    Sleep: number analyzed (Participants) | 15
    Sleep | 25.13 (5.33)
    Dexmedetomidine: number analyzed (Participants) | 20
    Dexmedetomidine | 22.95 (3.75)
    Ketamine: number analyzed (Participants) | 15
    Ketamine | 21.47 (3.14)
    Propofol: number analyzed (Participants) | 6
    Propofol | 22.83 (4.17)
    Midazolam: number analyzed (Participants) | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed for each row is the number of participants who completed that visit.
  Participants
    Total: Female | 7
    Total: Male | 20
    Sleep: number analyzed (Participants) | 15
    Sleep: Female | 4
    Sleep: Male | 11
    Dexmedetomidine: number analyzed (Participants) | 20
    Dexmedetomidine: Female | 6
    Dexmedetomidine: Male | 14
    Ketamine: number analyzed (Participants) | 15
    Ketamine: Female | 5
    Ketamine: Male | 10
    Propofol: number analyzed (Participants) | 6
    Propofol: Female | 2
    Propofol: Male | 4
    Midazolam: number analyzed (Participants) | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed for each row is the number of participants who completed that visit.
  Participants
    Total: Hispanic or Latino | 2
    Total: Not Hispanic or Latino | 17
    Total: Unknown or Not Reported | 8
    Sleep: number analyzed (Participants) | 15
    Sleep: Hispanic or Latino | 1
    Sleep: Not Hispanic or Latino | 6
    Sleep: Unknown or Not Reported | 8
    Dexmedetomidine: number analyzed (Participants) | 20
    Dexmedetomidine: Hispanic or Latino | 1
    Dexmedetomidine: Not Hispanic or Latino | 11
    Dexmedetomidine: Unknown or Not Reported | 8
    Ketamine: number analyzed (Participants) | 15
    Ketamine: Hispanic or Latino | 1
    Ketamine: Not Hispanic or Latino | 7
    Ketamine: Unknown or Not Reported | 7
    Propofol: number analyzed (Participants) | 6
    Propofol: Hispanic or Latino | 0
    Propofol: Not Hispanic or Latino | 2
    Propofol: Unknown or Not Reported | 4
    Midazolam: number analyzed (Participants) | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed for each row is the number of participants who completed that visit.
  Participants
    Total: American Indian or Alaska Native | 0
    Total: Asian | 1
    Total: Native Hawaiian or Other Pacific Islander | 1
    Total: Black or African American | 2
    Total: White | 15
    Total: More than one race | 0
    Total: Unknown or Not Reported | 8
    Sleep: number analyzed (Participants) | 15
    Sleep: American Indian or Alaska Native | 0
    Sleep: Asian | 1
    Sleep: Native Hawaiian or Other Pacific Islander | 1
    Sleep: Black or African American | 1
    Sleep: White | 4
    Sleep: More than one race | 0
    Sleep: Unknown or Not Reported | 8
    Dexmedetomidine: number analyzed (Participants) | 20
    Dexmedetomidine: American Indian or Alaska Native | 0
    Dexmedetomidine: Asian | 1
    Dexmedetomidine: Native Hawaiian or Other Pacific Islander | 0
    Dexmedetomidine: Black or African American | 1
    Dexmedetomidine: White | 10
    Dexmedetomidine: More than one race | 0
    Dexmedetomidine: Unknown or Not Reported | 8
    Ketamine: number analyzed (Participants) | 15
    Ketamine: American Indian or Alaska Native | 0
    Ketamine: Asian | 0
    Ketamine: Native Hawaiian or Other Pacific Islander | 0
    Ketamine: Black or African American | 0
    Ketamine: White | 8
    Ketamine: More than one race | 0
    Ketamine: Unknown or Not Reported | 7
    Propofol: number analyzed (Participants) | 6
    Propofol: American Indian or Alaska Native | 0
    Propofol: Asian | 0
    Propofol: Native Hawaiian or Other Pacific Islander | 0
    Propofol: Black or African American | 0
    Propofol: White | 2
    Propofol: More than one race | 0
    Propofol: Unknown or Not Reported | 4
    Midazolam: number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Occipital Delta Power Spectral Density by Conscious State and Study Group.
Description: The difference in spontaneous EEG slow wave activity over posterior cortex between states of consciousness measured with high-density EEG equipment and reported in spectral power in the delta band (1-4 Hz) at electrode Oz. Disconnected conscious experience (dreaming), connected conscious experience (awareness of the external world), and unconsciousness (no report) was assessed when participants were roused from sedation or sleep.
Time Frame: Intraoperative (During sedation-- up to 8 hours)
Population: No midazolam visit was ever conducted because no interested participants had reached that step of the drug sequence after it was added to the protocol in November of 2019.This was in large part due to the shutdown of in-person research activities in March of 2020 from the COVID-19 pandemic.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10(μV^2)
Groups:
- Dexmedetomidine: Standard drug visit activities: Participants were fitted with a saline gel EEG cap and a pre-sedation recording was collected. Participants' brain waves were recorded during rest, while responding to a standardized wake report form, and while performing a predictive coding cognitive task on a computer. Once the pre-sedation recording was collected, the faculty anesthesiologist began administering the study drug. A new EEG recording was started to monitor brain waves while all of the pre-sedation activities were repeated after the administration of the study drug.
  Dexmedetomidine-specific activities: Rapid infusion of 3.0 mg kg-1 h-1 was administered over a 10 min period followed by a 0.5 mg kg-1 h-1 maintenance infusion to achieve the first drug step. The second drug step was similarly achieved by a 10 min infusion of 3.0 mg kg-1 h-1 followed by a 1.5 mg kg-1 h-1 maintenance infusion. Duration of drug exposure was limited to 4 hours.
- Ketamine: Standard drug visit activities: Participants were fitted with a saline gel EEG cap and a pre-sedation recording was collected. Participants' brain waves were recorded during rest, while responding to a standardized wake report form, and while performing a predictive coding cognitive task on a computer. Once the pre-sedation recording was collected, the faculty anesthesiologist began administering the study drug. A new EEG recording was started to monitor brain waves while all of the pre-sedation activities were repeated after the administration of the study drug.
  Ketamine-specific activities: Ketamine was titrated using up to a 4.5mg/kg bolus over 10 minutes followed by 0.1-0.5mg/min intravenous infusion with 5 minutes between increments and titrated to desired observed alertness/sedation level. This infusion rate may be slowed further or stopped for patient safety concerns. Infusion rates will be adjusted using information from the target-controlled infusion model clinical judgment. Short-lived emergence delirium (confusion on awakening) may occur on emergence from ketamine anesthesia and this will be managed through standard clinical practice including administration of midazolam (up to 4mg IV) if required. Duration of drug exposure was limited to 4 hours.
- Propofol: Standard drug visit activities: Participants were fitted with a saline gel EEG cap and a pre-sedation recording was collected. Participants' brain waves were recorded during rest, while responding to a standardized wake report form, and while performing a predictive coding cognitive task on a computer. Once the pre-sedation recording was collected, the faculty anesthesiologist began administering the study drug. A new EEG recording was started to monitor brain waves while all of the pre-sedation activities were repeated after the administration of the study drug.
  Propofol-specific activities: A target-controlled infusion model used to predict plasma concentrations of propofol at 0.5 mcg/mL increments allowing 5-minutes to equilibrate between any step change. Dosing will be confined to FDA approved limits with up to a 2.5mg/kg bolus over 1 to 3 minute followed by an infusion of 50-200mcg/kg/min titrated to the desired observed alertness/sedation levels. Drug exposure was limited to 4 hours.
- Midazolam: Standard drug visit activities: Participants were fitted with a saline gel EEG cap and a pre-sedation recording was collected. Participants' brain waves were recorded during rest, while responding to a standardized wake report form, and while performing a predictive coding cognitive task on a computer. Once the pre-sedation recording was collected, the faculty anesthesiologist began administering the study drug. A new EEG recording was started to monitor brain waves while all of the pre-sedation activities were repeated after the administration of the study drug.
  Midazolam-specific activities: Initial boluses of up to 0.35mg/kg followed by doses up to 0.1mg/kg/h as a maintenance infusion. Duration of drug exposure was limited to 4 hours.
- Sleep: Participants were fitted with a saline gel EEG cap and a pre-sleep recording was collected. Participants' brain waves were recorded during rest, while responding to a standardized wake report form, and while performing a predictive coding cognitive task on a computer. After the pre-sleep recording, participants laid down within 30 minutes of their usual bedtime and were left to sleep for 2-3 hours. After this period, the participant was woken up every 15-30 minutes to answer standardized wake report form questions. After awaking a final time, the participant repeated 10 minutes of awake eyes open and eyes closed recordings as well as the predictive coding cognitive task on a computer.
Arm/Group | Dexmedetomidine | Ketamine | Propofol | Midazolam | Sleep
Number analyzed (Participants) | 20 | 15 | 6 | 0 | 15
log10(μV^2)
  Connected Consciousness | 2.37 [2.31 to 2.46] | 1.62 [1.57 to 1.68] | 2.05 [1.94 to 2.15] |  | 2.1 [2.03 to 2.18]
  Disconnected Consciousness | 2.57 [2.53 to 2.61] | 1.7 [1.57 to 1.84] | 2.34 [2.22 to 2.5] |  | 2.58 [2.52 to 2.65]
  Unconsciousness | 2.68 [2.61 to 2.75] | 1.46 [1.16 to 1.83] | 2.51 [2.31 to 2.68] |  | 2.63 [2.47 to 2.83]
Statistical Analysis 1: Comparison: Dexmedetomidine; Dexmedetomidine, Unconsciousness vs Disconnected Consciousness; Test type: Superiority; p = 0.012, Mixed Models Analysis — Statistical significance defined by p < 0.05; Slope = 0.110, Standard Error of Mean 0.043 — Estimate is a slope from a linear mixed effects model representing the difference in occipital delta power between unconsciousness and disconnected consciousness after adjusting for within-subject effects
Statistical Analysis 2: Comparison: Ketamine; Ketamine, Unconsciousness vs Disconnected Consciousness; Test type: Superiority; p = 0.236, Mixed Models Analysis — Statistical significance defined by p < 0.05; Slope = -0.238, Standard Error of Mean 0.199 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Propofol; Propofol, Unconsciousness vs Disconnected Consciousness; Test type: Superiority; p = 0.174, Mixed Models Analysis — Statistical significance defined by p < 0.05; Slope = 0.166, Standard Error of Mean 0.120 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Sleep; Sleep, Unconsciousness vs Disconnected Consciousness; Test type: Superiority; p = 0.640, Mixed Models Analysis — Statistical significance defined by p < 0.05; Slope = 0.052, Standard Error of Mean 0.111 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Instances of Disconnected Conscious Experience (Dreaming) vs Connected Conscious Experience (Awareness of External World).
Description: The number of instances of disconnected conscious experience (dreaming) versus connected conscious experience (awareness of the external world) during sedation is measured by subject self-report at the time of researcher initiated inquiry.
Time Frame: Intraoperative (During sedation-- up to 8 hours)
Population: There was no data collected for Midazolam or Sleep for this outcome measure.
Measure: Number; unit: number of instances
Arm/Group | Dexmedetomidine | Ketamine | Propofol | Midazolam | Sleep
Number analyzed (Participants) | 20 | 15 | 6 | 0 | 0
number of instances
  Instances of Connected Consciousness | 70 | 180 | 56 |  |
  Instances of Disconnected Consciousness | 226 | 30 | 22 |  |

3. Secondary Outcome: Effect of Study Drug on Ability to Correctly Identify Shapes/Images
Description: The ability to identify shapes/images in visual illusions measured by the NIH Toolbox. Will be reported by a computed score from NIH Toolbox for the Dimensional Change Card Sort Test (DCCS) and the Flanker Inhibitory Control & Attention Test (Flanker). Both Flanker and DCCS use a 2-vector scoring method that takes accuracy and reaction time (if accuracy >=80%) into account, resulting in a computed score that can range in value from 0-10. A higher score indicates better performance on the test.
Time Frame: Intraoperative (During sedation-- up to 8 hours)
Population: No data was collected for this outcome measure for Midazolam or Sleep
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine | Ketamine | Propofol | Midazolam | Sleep
Number analyzed (Participants) | 4 | 7 | 2 | 0 | 0
score on a scale
  Baseline NIH Toolbox Card Sorting Score | 8.83 (1.21) | 9.29 (0.59) | 9.45 (0.95) |  |
  Sedation NIH Toolbox Card Sorting Score | 7.85 (1.49) | 8.2 (0.99) | 6.94 (4.16) |  |
  Baseline NIH Toolbox Flanker Score | 9.14 (0.67) | 8.99 (0.83) | 9.48 (0.12) |  |
  Sedation NIH Toolbox Flanker Score | 6.62 (0.88) | 8.47 (0.93) | 8.36 (0.96) |  |
Statistical Analysis 1: Comparison: Dexmedetomidine; NIH Toolbox Card Sorting Score; Test type: Superiority; p = 0.134, t-test, 2 sided — Statistical significance defined by p < 0.05; 3 degrees of freedom
Statistical Analysis 2: Comparison: Ketamine; NIH Toolbox Card Sorting Score; Test type: Superiority; p = 0.012, t-test, 2 sided — Statistical significance defined by p < 0.05; 6 degrees of freedom
Statistical Analysis 3: Comparison: Propofol; NIH Toolbox Card Sorting Score; Test type: Superiority; p = 0.487, t-test, 2 sided — Statistical significance defined by p < 0.05; 1 degree of freedom
Statistical Analysis 4: Comparison: Dexmedetomidine; NIH Toolbox Flanker Score; Test type: Superiority; p = 0.046, t-test, 2 sided — Statistical significance defined by p < 0.05; 3 degrees of freedom
Statistical Analysis 5: Comparison: Ketamine; NIH Toolbox Flanker Score; Test type: Superiority; p = 0.010, t-test, 2 sided — Statistical significance defined by p < 0.05; 6 degrees of freedom
Statistical Analysis 6: Comparison: Propofol; NIH Toolbox Flanker Score; Test type: Superiority; p = 0.356, t-test, 2 sided — Statistical significance defined by p < 0.05

4. Secondary Outcome: Effect of Study Drug on Ability to Correctly Identify Images
Description: The ability to match sounds and images measured by the predictive coding task. Will be reported by a proportion correct as a decimal.
Time Frame: Intraoperative (During sedation-- up to 8 hours)
Population: No data was collected for this outcome measure for Midazolam or Sleep
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | Dexmedetomidine | Ketamine | Propofol | Midazolam | Sleep
Number analyzed (Participants) | 18 | 15 | 5 | 0 | 0
proportion correct
  Baseline Predictive Coding Task Accuracy | 0.916 (0.07) | 0.899 (0.07) | 0.91 (0.09) |  |
  Sedation Predictive Coding Task Accuracy | 0.793 (0.09) | 0.763 (0.1) | 0.734 (0.15) |  |
Statistical Analysis 1: Comparison: Dexmedetomidine; Predictive Coding Task Accuracy; Test type: Superiority; p < 0.001, t-test, 2 sided — Statistical significance defined by p < 0.05; 17 degrees of freedom
Statistical Analysis 2: Comparison: Ketamine; Predictive Coding Task Accuracy; Test type: Superiority; p < 0.001, t-test, 2 sided — Statistical significance defined by p < 0.05; 14 degrees of freedom
Statistical Analysis 3: Comparison: Propofol; Predictive Coding Task Accuracy; Test type: Superiority; p = 0.067, t-test, 2 sided — Statistical significance defined by p < 0.05; 4 degrees of freedom

5. Secondary Outcome: Effect of Study Drug on Ability to Form Implicit Memory
Description: Subjects will have a list of words read to them while under sedation and their ability to hear these words and form implicit memories of them will be assessed using a two-alternative forced choice task. Results will be reported as the average number of correct responses out of sixteen.
Time Frame: Intraoperative (During sedation-- up to 8 hours)
Population: There was no data collected for this outcome measure for Midazolam or Sleep.
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Dexmedetomidine | Ketamine | Propofol | Midazolam | Sleep
Number analyzed (Participants) | 18 | 12 | 5 | 0 | 0
correct responses | 8 (2.47) | 8.17 (1.70) | 9 (1.58) |  |
Statistical Analysis 1: Comparison: Dexmedetomidine; Null hypothesis is a 50% recall rate; Test type: Superiority; p = 0.5, t-test, 2 sided — Statistical significance defined by p < 0.05; 17 degrees of freedom
Statistical Analysis 2: Comparison: Ketamine; Null hypothesis is a 50% recall rate; Test type: Superiority; p = 0.37, t-test, 2 sided — Statistical significance defined by p < 0.05; 11 degrees of freedom
Statistical Analysis 3: Comparison: Propofol; Null hypothesis is a 50% recall rate; Test type: Superiority; p = 0.12, t-test, 2 sided — Statistical significance defined by p < 0.05; 4 degrees of freedom

ADVERSE EVENTS:
Time Frame: 24 hours after drug or sleep visit.
Description: Every participant was called by the study team the day after a drug or sleep visit and asked to report any adverse events experienced since the visit. If any reported, study team reported them to study physician, and completed a serious adverse event tracking log if needed. If the adverse event fulfilled criteria outlined in protocol, it would be reported to the internal review board at UW- Madison.
Arm/Group | Dexmedetomidine | Ketamine | Propofol | Midazolam | Sleep
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/15 | 0/6 | 0/0 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/15 | 0/6 | 0/0 | 0/15
Other Adverse Events (participants affected / at risk) | 5/20 | 6/15 | 1/6 | 0/0 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=20) | Ketamine (N=15) | Propofol (N=6) | Midazolam (N=0) | Sleep (N=15)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Mild Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The fourth study drug was changed from sevoflurane to midazolam in November of 2019 due to concerns about conducting experiments in patients inhaling a volatile anesthetic through a face mask and the difficulty we would have with communicating with patients. The cessation of human subjects research due to the COVID-19 pandemic and amended institutional guidelines for conducting in-person research caused far fewer participants to be recruited than was planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03284307/Prot_SAP_002.pdf
  • Informed Consent Form (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03284307/ICF_001.pdf